CLINICAL TRIAL: NCT00803946
Title: A Randomized, Single-Dose, Two-Way Crossover Relative Bioavailability Study of Ibuprofen Tablet Formulations in Normal, Healthy Men and Women Following Standard Meal
Brief Title: Bioequivalence Study Between Two Oral Formulations of Ibuprofen 800 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Perrigo Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30275
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Bioequivalency
Keywords: bioequivalency; ibuprofen
MeSH Terms: interventions — Ibuprofen

ARMS (2):
- Test Product (Active Comparator)
  Interventions: Drug: Ibuprofen Tablets, 800 mg
- Reference Product (Active Comparator)
  Interventions: Drug: Ibuprofen Tablets, 800 mg

INTERVENTIONS:
Drug: Ibuprofen Tablets, 800 mg

SUMMARY:
Compare the rate and extent of absorption of two oral formulations of Ibuprofen 800 mg Tablets, administered as a 1 x 800 mg tablet, under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women, 18 years of age or older
* body mass index between 19 and 30
* willing to participate and sign a copy of the informed consent form

Exclusion Criteria:

* history of allergy or hypersensitivity to ibuprofen
* recent history of drug or alcohol addiction or abuse
* pregnant or lactating women
* use of tobacco products during the past 3 months
* evidence of a clinically significant disorder or whose laboratory results were deemed to be clinically significant
* receipt of any drugs as part of a research study within 30 days prior to study dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-11; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence was assessed on the pharmacokinetic variables Cmax, AUC,0-t, and AUC,0-infinity